CLINICAL TRIAL: NCT04373239
Title: Trends in Live Birth Rates Attributable to Assisted Reproductive Technology in British Columbia
Status: Completed | Type: Observational
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Mohamed Bedaiwy, Principle Investigator, University of British Columbia
Other Study IDs: H20-00461-B
Record Dates: First submitted 2020-04-29; First posted 2020-05-04 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2020-04

CONDITIONS: Assisted Reproductive Techniques
MeSH Terms: interventions — Reproductive Techniques, Assisted

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Women in BC conceiving by ART: All women in BC registered in the Perinatal Services BC database having undergone Assisted Reproductive Technology. Assisted Reproductive Technology will consist of in vitro fertilization (+/-ICSI). Data from April 1, 2008 to March 31 2018 will be analyzed for live birth rate.
  Interventions: Procedure: Assisted Reproductive Technology
- Women in BC conceiving spontaneously: he comparison group will be all women in BC registered in the Perinatal Services BC database with spontaneously conceived pregnancies between April 1, 2008 to March 31 2018.

INTERVENTIONS:
Procedure: Assisted Reproductive Technology — Assisted reproductive technology includes IVF and IVF+ICSI.
  Groups: Women in BC conceiving by ART

SUMMARY:
Investigators will examine trends in ART use in BC specifically. The use of ART has drastically changed the management of infertility, with worldwide estimates exceeding 1.8 million ART cycles in 2010 alone. Moreover, an excess of six million children have been conceived using ART. Although various countries have published their live birth rates associated with common ART treatment strategies, British Columbia has yet report on its rates. With varying differences in ART practices, whether clinical or laboratory, it is expected live birth rates due to ART to vary depending on region analyzed. Analyzing the live birth rate in BC would not only allow for a benchmark for assessing future improvement, and trends in infertility diagnosis and management, but also allow for comparison to other provinces and countries. The aim of this part of the study is to describe ART cycle contribution to live birth rate in BC from April 2008 to March 2018, which has not been addressed in the literature as of yet. Not only will it give healthcare providers and patients information about this emerging approach to infertility but also provide a impetus for healthy policy makers to adopt a model for partially or fully publicly funded ART, as seen in Ontario and soon Quebec.

DETAILED DESCRIPTION:
Perinatal Services BC maintains a current database on live births, antepartum, intrapartum and postpartum outcomes; including details of ART if used to conceive. Live birth rate, for the purposes of this study, will be defined as the birth of at least one live born baby, with the birth of twins or higher order multiples considered as one live birth. The birth rate for ART will be taken as a proportion for birth rate from ART over total birth rate for given calendar year and the overall period of analysis. Data from April 1 2008 to March 31 2018 on autologous ART treatment cycles and outcomes will be extracted from this database, with approval. Overall proportion of ART contributing to live birth rate will be analyzed as well as sub categorical analysis based on age (younger than 30, 30-34 years, 35-39 years, 40-44 years, and 45 years and older). Only nulliparous women will be included in this study.

Moreover, data will be analyzed by calendar year in which baby from ART delivered to evaluate overall trends in ART outcomes. The total live birth rate for all of BC will serve as the denominator.

Although the data will be reviewed and rules interpreted by the principal investigator of this study, a biostatistician will be hired to carry out the necessary statistical analysis.

ELIGIBILITY:
Inclusion Criteria:

* Nulliparous women registered in Perinatal Services BC database with live birth between April 2008 and March 2018

Exclusion Criteria:

* multiparous women
* women with missing data in Perinatal Services BC database including gravid, parity, age, date of birth

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All women registered in Perinatal Services BC database with live births between April 2008 and March 2018.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2008-04 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Live birth rate | Date of delivery
  Live birth rate

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Bedaiwy, MD, PhD, Principal Investigator — University of British Columbia

IPD SHARING:
Plan to Share IPD: No